CLINICAL TRIAL: NCT03024853
Title: Efficacy of Different Versions of the Best Possible Self Intervention: a Randomized Controlled Trial
Brief Title: Efficacy of Different Versions of the Best Possible Self Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, Full Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1415802387094
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: General Population
Keywords: Best Possible Self; Positive Intervention; Optimism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- BPS PAST (Experimental): Participants write down about themselves in a past when they displayed their best self. Then, they make a video with this text and a chosen song, watch the video and then they visualize (imagine) the content.
  Interventions: Behavioral: BPS PAST
- BPS PRESENT (Experimental): Participants write down about themselves in in the present, focusing on what currently makes the best version of themselves (skills, features...). Then, they make a video with this text and a chosen song, watch the video and then they visualize (imagine) the content.
  Interventions: Behavioral: BPS PRESENT
- BPS FUTURE (Experimental): Participants write down about themselves in the future after everything has gone as well as it possibly could. Then, they make a video with this text and a chosen song, watch the video and then they visualize (imagine) the content.
  This is the original BPS exercise (already validated in other studies).
  Interventions: Behavioral: BPS FUTURE
- CONTROL (Active Comparator): Participants write down the activities they did during the last 24 hours. Then, they visualize (imagine) the content. They practice the visualization exercise for 7 consecutive days.
  Interventions: Behavioral: CONTROL

INTERVENTIONS:
Behavioral: BPS PAST
  Arms: BPS PAST
Behavioral: BPS PRESENT
  Arms: BPS PRESENT
Behavioral: BPS FUTURE
  Arms: BPS FUTURE
Behavioral: CONTROL
  Arms: CONTROL

SUMMARY:
The aim of this study is to analyze the efficacy of several variations of an already validated Positive Psychology Intervention (PPI) called Best Possible Self, using Information and Communication Technologies (ICT) in general population. Participants are randomly assigned to one of 4 conditions: BPS PAST condition, BPS PRESENT condition, BPS FUTURE condition, and CONTROL condition (daily activities).

DETAILED DESCRIPTION:
Intervention lasts 7 days. Participants come to the laboratory the first day, they fill up assessment questionnaires and practice the assigned exercise. Then, they practice the assigned exercise for 6 more days at home.

The main hypothesis is that all three experimental conditions will enhance wellbeing comparing to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years old or older.
* Participants must be willing to participate in the study.
* Participants must have computer with Internet access and e-mail address.

Exclusion Criteria:

* To suffer from moderated or severe depression as established by a score of 20 or more in the Beck Inventory of Depression (BDI-II; Beck, 1996).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change from Positive and Negative Affect Scale (PANAS; Watson, Clark & Tellegen, 1988; Sandín et al., 1999) from baseline to post-in | Change from pre-intervention to post-intervention (1 week) and follow-up (1 month, 3 months).

SECONDARY OUTCOMES:
New General Self-Efficacy Scale (NGSES; Chen, Gully & Eden, 2001) | Change from pre-intervention to post-intervention (1 week) and follow-up (1 month, 3 months).
Life Orientation Test (LOT-R; Otero, Luengo, Romero Gómez & Castro, 1998; Scheier, Carver & Bridges, 1994). | Change from pre-intervention to post-intervention (1 week) and follow-up (1 month, 3 months).
Fordyce Happiness Scale (Fordyce, 1988) | Change from pre-intervention to post-intervention (1 week) and follow-up (1 month, 3 months).
Temporal Satisfaction with Life Scale (TSWLS; Pavot, Diener & Suh, 1998) | Change from pre-intervention to post-intervention (1 week) and follow-up (1 month, 3 months).

OTHER OUTCOMES:
Self-Concordant Motivation (SCM; Sheldon & Elliot, 1999) | Day 1
  This scale measures the intrinsic motivation of participants' when practicing the assigned activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Baños, Professor, Study Director — University of Valencia; Ernestina Etchemendy, Researcher, Study Director — University of Teruel; Alba Carrillo, PhD student, Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] King L. The Health Benefits of Writing About Life Goals. Personality and Social Psychology Bulletin 27(7): 798-807, 2001.
- [Background] Sheldon KM, Lyubomirsky S. How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology 1(2): 73-82, 2006.
- [Background] Peters ML, Flink IK, Boersma K, Linton SJ. Manipulating optimism: Can imagining a best possible self be used to increase positive future expectancies? The Journal of Positive Psychology 5(3): 204-211, 2010.